CLINICAL TRIAL: NCT00824044
Title: QEEG Predictors of Response for Psychotherapy Compared to Pharmacotherapy in Depression
Brief Title: Quantitative Electroencephalogram (QEEG) Predictors of Response to Psychotherapy Versus Antidepressant Treatment in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Amy Farabaugh, PhD, Staff psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2008-P-000838
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder (MDD); Cognitive Behavioral Therapy (CBT); Escitalopram; Quantitative EEG (QEEG)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Escitalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Active Comparator): CBT is a manualized therapeutic treatment for depression based on principles of cognitive restructuring and behavioral changes.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Escitalopram (Active Comparator): Escitalopram or Lexapro is a Selective Serotonin Reuptake Inhibitor (SSRI) used to treat depression
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The CBT group will receive weekly 50-minute individual sessions over the course of 12 weeks conducted by experienced therapists who are trained in manual based CBT.
  Arms: Cognitive Behavioral Therapy (CBT)
Drug: Escitalopram — The medication group will receive open label treatment of escitalopram, 10-20 mg/day, flexible dose, for 12 weeks, and will be seen every two weeks by a study physician.
  Other Names: Lexapro
  Arms: Escitalopram

SUMMARY:
The purpose of this research study is to find out if a test can predict whether someone with depression will get better with treatment. We also want to find out whether there are changes in the brains of depressed patients having different types of treatment (drug therapy vs. talk therapy). We hope that a test called QEEG (Quantitative Electroencephalogram) can tell us if a treatment is going to work, even before the person starts to feel better.

Hypothesis 1: Response to treatment will correlate with changes in QEEG metrics.

Hypothesis 2: QEEG parameters, different from those that predict response to pharmacotherapy, will be associated with response to CBT.

DETAILED DESCRIPTION:
To our knowledge, QEEG has not been studied in the prediction of response to CBT, an important and widely used non-pharmacologic approach to treating depression. Establishing QEEG technology as a predictor of response to CBT could help to guide treatment selection for individual patients. It is probable that certain patient populations are more likely to respond to either psychotherapeutic or psychopharmacological interventions, while others may benefit from a combination of treatment modalities. This study will provide preliminary information about the utility of QEEG as a predictor of response in psychotherapy and will furnish the knowledge base of QEEG changes related to clinical variables, providing pilot data for a study in a larger sample. We have hypothesized that clinical response will correlate with changes in QEEG metrics from beginning to two weeks after treatment, and that QEEG parameters, different from those that predict response to pharmacotherapy, will be associated with response to CBT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be adults, ages 18 to 75 years.
* Written informed consent
* MDD, current according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV)
* 17-item Hamilton Depression Rating Scale (HAM-D-17) score of > 14 at baseline.
* Subjects who are not currently taking any antidepressant or other psychotropic medications and who have been free of these medications for 4 weeks prior to screening visit.

Exclusion Criteria:

* Women who are pregnant, lactating, or planning a pregnancy during the study.
* Women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or a partner with vasectomy).
* Any uncontrolled psychiatric disorder.
* Current use of psychotropic medications.
* Psychotic features in the current episode or a history of psychotic features.
* Alcohol or substance abuse or dependence within the past three months.
* History of head trauma or seizure disorder.
* History of intolerance of the study medication.
* Failure to respond to escitalopram up to 20 mg for at least 6 weeks.
* Failure to respond to 2 or more adequate antidepressant trials (6 weeks or longer on a therapeutic dose, equivalent to fluoxetine 40mg) in the current episode.
* Currently enrolled in other depression-focused psychotherapy and unwilling to cease treatment.
* Subjects who, per clinical judgment, are not appropriate candidates for CBT or SSRIs.
* History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, including alcohol, active within the last 3 months.
* Serious suicide or homicide risk, as assessed by the evaluating clinician or a score of 4 on the third item of the HAM-D.
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Farabaugh, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was screened on January 6, 2009, and the last patient was screened on October 26, 2010. The study was completed at the Depression Clinical and Research Program at Massachusetts General Hospital.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) | Escitalopram
Started | 23 | 16
Completed | 14 | 10
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) | Escitalopram | Total
Number analyzed (Participants) | 23 | 16 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data unavailable for 2 participants
  years
    number analyzed (Participants) | 22 | 15 | 37
    (all) | 44.8 (14.2) | 43.3 (15.5) | 43.9 (14.8)
Age, Customized [Number; unit: participants] — Age at screen was not available for 2 participants.
  participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 19 | 14 | 33
    >=65 years | 3 | 1 | 4
    Age unknown | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 11 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 23 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAM-D-17) Scores
Description: The Hamilton Depression Rating Scale is a clinician-rated scale used to rate depression severity. The maximum score is a 50 and the minimum score is a 0, where higher scores indicate greater severity. Scores from 14 to 18 indicate moderately severe depression.
Time Frame: 12 weeks
Population: The number of participants for analysis was based on the number of participants who completed treatment (12 weeks of CBT or medication)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy (CBT): Patients receive twelve weekly 50-minute individual sessions of cognitive-behavioral therapy over the course of twelve weeks. Scores on the HAM-D-17 at Week 12 are the primary outcome measure.
- Escitalopram: Patients received 10-20 mg/day of flexible-dose open-label escitalopram for 12 weeks. Scores on the HAM-D-17 at Week 12 are the primary outcome measure.
Arm/Group | Cognitive Behavioral Therapy (CBT) | Escitalopram
Number analyzed (Participants) | 14 | 9
units on a scale | 10.64 (6.44) | 13.78 (9.40)

2. Primary Outcome: Change in Absolute Beta Power in Channel 4
Description: Change between baseline and LOCF in absolute power of the beta wave recorded from channel 4 of the EEG
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Groups:
- Non Responders in CBT Arm: Individuals randomized to the CBT group who did not respond to the CBT treatment. Response defined as greater than 50% reduction in HAM D scores
- Responders in CBT Arm: Individuals randomized to the CBT group who did respond to the CBT treatment. Response defined as greater than 50% reduction in HAM D scores
- Non Responders in Medication Arm: Individuals randomized to the CBT group who did not respond to the Medication treatment. Response defined as greater than 50% reduction in HAM D scores
- Responders in Medication Arm: Individuals randomized to the medication group who did respond to the medication treatment. Response defined as greater than 50% reduction in HAM D scores
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0930 (.13602) | -.0102 (.09301) | .0683 (.151) | .0056 (.1084)

3. Primary Outcome: Change in Absolute Theta Power From Channel 1
Description: Change between baseline and LOCF in relative power of the theta wave recorded from channel 1 of the EEG. Relative power refers to the percentage of power in the theta wave compared with the total power in the patient's EEG.
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .225 (.02765) | -.0455 (.07683) | .0075 (.0734) | .003 (.0535)

4. Primary Outcome: Change in Relative Theta Power Channel 3
Description: Change between baseline and LOCF in relative power of the theta wave recorded from channel 3 of the EEG. Relative power refers to the percentage of power in the theta wave compared with the total power in the patient's EEG.
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0362 (.04460) | -.0090 (.0859) | .0015 (.02993) | .272 (.06577)

5. Primary Outcome: Change in Relative Theta Power From Channel 4
Description: Change between baseline and LOCF in relative power of the theta wave recorded from channel 4 of the EEG. Relative power refers to the percentage of power in the theta wave compared with the total power in the patient's EEG.
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0336 (.04428) | -.0009 (.03210) | .0076 (.03678) | .0070 (.04429)

6. Primary Outcome: Change in Relative Beta Power From Channel 4
Description: Change between baseline and LOCF in relative power of the beetawave recorded from channel 4 of the EEG. Relative power refers to the percentage of power in the beta wave compared with the total power in the patient's EEG.
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0483 (.03560) | .0173 (.02921) | .0063 (.03758) | .0179 (.02929)

7. Primary Outcome: Change in Absolute Beta Power From the Ear Channel
Description: Change between baseline and LOCF in absolute power of the beta wave recorded from the ear channel of the EEG. The ear channel refers to the average of channels 3 and 4.
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0537 (.08943) | -.0167 (.07461) | .0670 (.14412) | -.01401 (.08307)

8. Primary Outcome: Change in Relative Theta Power From Temporal Channel
Description: Change between baseline and LOCF in relative power of the theta wave recorded from the temporal channel of the EEG. Relative power refers to the percentage of power in the theta wave compared with the total power in the patient's EEG. The temporal channel refers to the average of channels 1 and 2
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0182 (.02003) | -.0159 (.03422) | .0125 (.07914) | .0027 (.03688)

9. Primary Outcome: Change in Relative Theta Power From Ear Channel
Description: Change between baseline and LOCF in relative power of the theta wave recorded from the ear channel of the EEG. Relative power refers to the percentage of power in the theta wave compared with the total power in the patient's EEG. The ear channel refers to the average of channels 3 and 4
Time Frame: 12 weeks
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
Hz | .0349 (.04440) | -.0050 (.03487) | .0046 (.02858) | .0171 (.04103)

10. Primary Outcome: Percent Change in Relative Theta Power From Week 1 of the Ear Channel
Description: Percent change between baseline and week 1 in relative power of the theta wave recorded from the ear channel of the EEG. Relative power refers to the percentage of power in the theta wave compared with the total power in the patient's EEG. The ear channel refers to the average of channels 3 and 4
Time Frame: 1 week
Population: EEG data only available for 11 participants from CBT arm and 11 participants from Medication arm
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Non Responders in CBT Arm | Responders in CBT Arm | Non Responders in Medication Arm | Responders in Medication Arm
Number analyzed (Participants) | 5 | 6 | 5 | 6
percent | 44.1809 (42.17256) | 8 (27.45993) | 7.5180 (29.37028) | 23.3718 (41.25936)

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Therapy (CBT) | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/16
Other Adverse Events (participants affected / at risk) | 0/23 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (CBT) (N=23) | Escitalopram (N=16)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) — 2/16 participants reported nausea
Headache (General disorders) | 0 (0) | 4 (5) — 4/16 participants reported experiencing headaches.
syncopal episode (Nervous system disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 0 (0) | 1 (1)
dry mouth (General disorders) | 0 (0) | 3 (3)
irregular menses (Reproductive system and breast disorders) | 0 (0) | 1 (1)
knee aching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
migraines (General disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
sedation (General disorders) | 0 (0) | 1 (1)
sweatiness (General disorders) | 0 (0) | 2 (2)
sleepiness (General disorders) | 0 (0) | 2 (3)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
fidgetiness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2009-11-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT00824044/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT00824044/SAP_001.pdf